CLINICAL TRIAL: NCT02782845
Title: Expanded Access Program of Pegfilgrastim in Patients With Non-Hodgkin Lymphoma (NHL)
Brief Title: An Expanded Access Program of Pegfilgrastim (Neulastim) in Participants With Non-Hodgkin's Lymphoma (NHL)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML19812
Record Dates: First submitted 2016-05-16; First posted 2016-05-25 (Estimated); Last update posted 2016-11-21 (Estimated); Status verified 2016-09

CONDITIONS: Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Drug Therapy; pegfilgrastim

ARMS (1):
- Pegfilgrastim (Experimental): Participants will receive CT or ICT for 6 cycles on Days 1-6, as per standard of care. Protocol does not specify any choice of CT or ICT drugs. Participants will receive pegfilgrastim at a fixed dose of 6 mg subcutaneously, 24 hours after the last dose of CT or ICT in each treatment cycle. CT or ICT cycles of 21 days, as per standard of care.
  Interventions: Drug: Chemotherapy; Drug: Immunochemotherapy; Drug: Pegfilgrastim

INTERVENTIONS:
Drug: Chemotherapy — The choice of CT will be as per standard of care and protocol does not specify any particular CT drug.
Drug: Immunochemotherapy — The choice of ICT will be as per standard of care and protocol does not specify any particular ICT drug.
Drug: Pegfilgrastim — Pegfilgrastim will be administered at a fixed dose of 6 mg subcutaneously 24 hours after the last dose of CT or ICT is received for 6 cycles.
  Other Names: Neulastim

SUMMARY:
This study will assess the prophylactic effect of pegfilgrastim (Neulastim) on febrile and/or Grade IV neutropenia in participants receiving chemotherapy (CT) or immunochemotherapy (ICT) as first or second line treatment for NHL. Pegfilgrastim will be administered at a fixed dose of 6 milligrams (mg) subcutaneously 24 hours after the last dose of CT or ICT in each treatment cycle.

ELIGIBILITY:
Inclusion Criteria:

* NHL supported by an Immunohistochemical report
* Eastern Cooperative Oncology Group (ECOG) performance status greater than or equal to (>/=) 2
* Total serum bilirubin less than (<) 2 times upper limit of normal (ULN)
* Absolute neutrophil count (ANC) greater than (>) 2 x10^9 per liter (/L)

Exclusion Criteria:

* Bone marrow compromised > 10 percent (%)
* Any malignant myeloid condition
* Active infections requiring systemic anti-infectious therapies (antibiotics, antifungal drugs, antiviral drugs) within 72 hours prior to CT or ICT initiation
* Known hypersensitivity reactions to Escherichia coli derived products
* Pregnant or nursing participants. Women with childbearing potential should use a safe contraceptive method

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2006-06; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Febrile Neutropenia (Absolute Neutrophil Count [ANC] <0.5x10^9/L and Temperature ≥38 degrees Celsius) And/Or Grade IV Neutropenia (ANC<0.5x10^9/L) in Cycle 1 | Cycle 1 (Up to 21 days)

SECONDARY OUTCOMES:
Percentage of Participants with Febrile Neutropenia (ANC <0.5x10^9/L and temperature ≥38 degrees Celsius) And/Or Grade IV Neutropenia (ANC<0.5x10^9/L) in Cycles 2 to 6 | Cycles 2 to 6 (Up to 105 days)
Percentage of Participants with Adverse Events | up to approximately 1.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (12):
- Bogotá, Colombia
- Mexico (11):
  - Chihuahua City
  - Estado de México
  - Guadalajara
  - León
  - Mexico City
  - Obregón
  - Puebla City
  - Querétaro
  - Tepic
  - Toluca
  - Veracruz